CLINICAL TRIAL: NCT02304471
Title: Circulating Long Non-coding RNAs and Cardiovascular Morbidities in Chronic Kidney Disease and End-Stage Renal Disease
Brief Title: Circulating lncRNA and CV Morbidities in CKD and ESRD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201409019RINB
Record Dates: First submitted 2014-11-26; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Kidney Disease; End-stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: healthy subjects
- CKD: chronic kidney disease
- ESRD: end-stage renal disease

SUMMARY:
Cardiovascular disease is the major cause of morbidity and death in patients with chronic kidney disease (CKD) and end-stage renal disease (ESRD). The mechanisms linking impaired renal function and increased risk for cardiovascular diseases, however, remain elusive.

Long non-coding RNAs (lncRNAs) is a heterogeneous group of non-coding transcripts longer than 200 nucleotides. While the roles of lncRNAs in human diseases including cancer and neurodegenerative disorders are beginning to emerge, it remains unclear how lncRNA regulation contributes to cardiovascular complications in patients with renal dysfunction.

In this proposal, the investigators seek to apply next-generation sequencing technology to investigate circulating lncRNA expression in control subjects and in patients with CKD and ESRD. The investigators will test the hypothesis that circulating lncRNA expression signature can reflect the underlying kidney disease states in patients with CKD and ESRD. A gene co-expression network analysis will be conducted to identify lncRNAs that are functionally involved in the pathogenesis of CKD and ESRD. Next, the investigators will identify circulating lncRNAs that are indicative of cardiovascular dysfunction in ESRD patients. Finally, the investigators propose to test the hypothesis that circulating lncRNAs can be novel prognostic biomarkers to predict cardiovascular outcomes and renal function progression in CKD patients. The results from these experiments will lead to better understanding of how circulating lncRNAs contribute to uremic cardiovascular complications and renal function progression.

DETAILED DESCRIPTION:
Cardiovascular disease is the major cause of morbidity and death in patients with chronic kidney disease (CKD) and end-stage renal disease (ESRD). Patients with CKD and ESRD are at high risk for myocardial dysfunction, ischemia and heart failure. The mechanisms linking impaired renal function and increased risk for cardiovascular diseases, however, remain elusive. In addition, conventional therapeutics proven effective in reducing cardiovascular events in general population fail to provide similar benefits in uremic patients. There is a clear need to identify novel mediators of cardiovascular complications in uremic patients to provide insights into the pathogenesis, to tailor clinical care based on cardiovascular risks, and to develop new therapeutic strategies.

It has become increasingly clear that the transcription of the eukaryotic genome is far more pervasive and complex than previously appreciated. While the expression of messenger RNAs (mRNAs) and microRNAs (miRNAs) account for only ~1% of all transcribed species, up to 90% of the mammalian genome is transcribed as long non-coding RNAs (lncRNAs), a heterogeneous group of non-coding transcripts longer than 200 nucleotides. LncRNAs have been shown to be functional and involved in specific physiological and pathological processes through epigenetic, transcriptional and post-transcriptional mechanisms. While the roles of lncRNAs in human diseases including cancer and neurodegenerative disorders are beginning to emerge, it remains unclear how lncRNA regulation contributes to cardiovascular complications in patients with renal dysfunction.

In this proposal, we seek to apply next-generation sequencing technology to investigate circulating (plasma and peripheral blood mononuclear cells [PBMC]) lncRNA expression in control subjects and in patients with CKD and ESRD. We will test the hypothesis that circulating lncRNA expression signature can reflect the underlying kidney disease states in patients with CKD and ESRD. A gene co-expression network analysis will be conducted to identify lncRNAs that are functionally involved in the pathogenesis of CKD and ESRD. Next, we will identify circulating lncRNAs that are indicative of cardiovascular dysfunction in ESRD patients. The hypothesis that circulating lncRNAs can be used to predict the progression of myocardial dysfunction, the occurrence of adverse cardiovascular events and death among patients with ESRD, will be tested. The sensitivity and specificity of using circulating lncRNAs to predict cardiovascular function/outcomes in ESRD patients will be tested prospectively in an independent ESRD population. Finally, we propose to test the hypothesis that circulating lncRNAs can be novel prognostic biomarkers to predict cardiovascular outcomes and renal function progression in CKD patients. The results from these experiments will lead to better understanding of how circulating lncRNAs contribute to uremic cardiovascular complications and renal function progression. These experiments will also help to design better diagnostic and prognostic tools in CKD/ESRD patients, as well as to develop novel therapeutic strategies to treat or prevent CKD progression and uremic cardiovascular complications.

ELIGIBILITY:
Inclusion Criteria:

* 1.Adult patients with various stages 1-5 of CKD will be enrolled at outpatient clinic. Definition and staging of CKD were defined by estimated glomerular filtration rate by the Modification of Diet in Renal Disease study equation.
* 2.Patients with ESRD under maintenance hemodialysis or peritoneal dialysis will also be included.

Exclusion Criteria:

* 1.age younger than 20 years or older than 80 years.
* 2.pregnant woman.
* 3.patients already received kidney transplantation.
* 4.recent hospitalization within previous one month.
* 5.for ESRD patients, receiving maintenance hemodialysis or peritoneal dialysis for less than 3 months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD, ESRD, Healthy controls
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Adverse cardiovascular events (acute myocardial ischemia, life-threatening atrial/ventricular arrhythmias, acute decompensated heart failure, stroke and cardiovascular death) | 3 years
  Adverse cardiovascular events including acute myocardial ischemia, life-threatening atrial/ventricular arrhythmias, acute decompensated heart failure, stroke and cardiovascular death will be recorded over the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Fu Lai, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan